CLINICAL TRIAL: NCT04625894
Title: Phase I Clinical Trial of Multisite Stereotactic Ablative Radiotherapy (SABR) Combined With Camrelizumab in Patients With Oligometastatic Gastrointestinal Cancer
Brief Title: The Combination of Immunotherapy and Stereotactic Ablative Radiotherapy in Oligometastatic Gastrointestinal Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhen Zhang, Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MA-CRC-I-002
Record Dates: First submitted 2020-11-06; First posted 2020-11-12 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: Oligometastatic Gastrointestinal Cancer
MeSH Terms: interventions — camrelizumab; Injections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental): Patients with oligometastatic gastrointestinal cancer will receive multisite SABR, followed by Camrelizumab within one week from completion of radiation. Camrelizumab for injection at 200 mg, d1, q2w, 14-day cycle will continue for up to two years until disease progression, unacceptable toxicity or patient withdrawal.
  Interventions: Radiation: Stereotactic Ablative Radiotherapy (SABR); Drug: Camrelizumab for injection (200 mg, iv), D1, Q2W, 14-day cycle

INTERVENTIONS:
Radiation: Stereotactic Ablative Radiotherapy (SABR) — To irradiate as many metastatic lesions as possible, in the precondition that normal tissues can tolerate. Target dose will be adjusted depending on site of the lesion and organs at risk (BED > 100Gy). Sequence of irradiation for multiple metastases will be at the discretion of the investigators based on their experience.
Drug: Camrelizumab for injection (200 mg, iv), D1, Q2W, 14-day cycle — Administration of Carrelizumab will be started within one week upon SABR completion, and will be continued for up to two years until disease progression, unacceptable toxicity or patient withdrawal.

SUMMARY:
This is a single-center, open-label, single-arm phase I clinical study to exploratory observe and evaluate the efficacy and safety of anti-PD-1 antibody (Camrelizumab for Injection) combined with multisite stereotactic ablative radiotherapy (SABR) in patients with oligometastatic gastrointestinal cancer.

According to the origin site of metastases, this study will consist of three subgroups, including gastric carcinoma group, colorectal carcinoma group and hepatocellular carcinoma group. For each of the subgroup, seven eligible patients with oligometastatic cancer originating from stomach, colon and liver, respectively will be recruited. All patients will receive multisite SABR followed by immunotherapy of Camrelizumab within one week from completion. Camrelizumab will be administered at a fixed dose of 200 mg intravenously (iv) on D1 in a 14-day cycle. The treatment will continue for up to two years until disease progression, unacceptable toxicity or patient withdrawal.

Tumor tissue samples, sections, paraffin blocks or biopsy blocks, and biomarkers, including but not limited to PD-L1 expression level and the proportion of positive cells, TMB level and MMR status, will be collected from subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-70 years old, regardless of gender;
2. Fully informed and willing to provide written informed consent for the trial;
3. ECOG performance status 0-1;
4. Expected survival time ≥ 6 months;
5. Has gastric carcinoma /colorectal carcinoma / hepatocellular carcinoma, confirmed by histopathology (or pathology consultation in our hospital) and measurable oligometastatic lesions on imaging (RECIST version 1.1); pathological diagnosis confirmation of oligometastatic lesions using biopsy tissue samples (e.g. obtained by hollow core needle, biopsy, excision, etc.) is recommended but not required;
6. Has undergone curative treatment on the primary lesion at least three months ago, without local progression;
7. Has received standard treatment prior to enrolment, except for any type of immunotherapy;
8. Has no more than three metastatic lesions detected on imaging in single organ (e.g. lung, liver, brain, bone, etc.), and the total number of metastases is no more than five;
9. Multiple sites of lesions can be safely treated by SABR; and the maximum diameter of each lesion for irradiation is no more than 5cm.
10. Contraindicated for surgery or the participant refuses to receive surgery.
11. Has adequate organ function to tolerate the regimen:
12. Bone marrow function: neutrophils ≥ 1.5 × 109/L, platelets ≥ 100 × 109/L, hemoglobin ≥ 90 g/L;
13. Liver and kidney function: serum creatinine ≤ 1.5 times the upper limit of normal; AST and ALT ≤ 2.5 times the upper limit of normal or the presence of liver metastasis ≤ 5 times the upper limit of normal; total bilirubin ≤ 1.5 times the upper limit of normal, or patients with Gilbert's syndrome ≤ 2.5 times the upper limit of normal;
14. Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up
15. Non-lactating patients.

Exclusion Criteria:

1. Pregnant or lactating women
2. Serious medical comorbidities precluding radiotherapy
3. Prior radiotherapy to a site requiring treatment
4. Malignant pleural effusion
5. Inability to treat all sites of active disease
6. Has clinical or radiologic evidence of spinal cord compression or tumor within 3mm of spinal cord on MRI.
7. Dominant brain metastasis requiring surgical decompression
8. Has prior treatment with cancer immunotherapy including, but not limited to immune checkpoint inhibitors.
9. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy at a dose of >10 mg Prednisone daily or equivalent at time of trial treatment.
10. Has a known history of active Bacillus Tuberculosis
11. Has active autoimmune disease that has required systemic treatment in the past 2 years
12. Hypersensitivity to PD-1 inhibitor or any of its excipients.
13. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study day 1 or who has not recovered from adverse events due to a previously administered agent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2020-12 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicities (DLT) | Up to 2 years
  Defined as treatment-related Grade 3 or higher toxicities (excluding asymptomatic biochemical abnormalities) within 3 months, starting from the first day of radiotherapy. Toxicities will be assessed and graded according to NCI-CTCAE v5.0.

SECONDARY OUTCOMES:
Adverse events (AEs) | Up to 2 years
  Assessed according to NCI-CTCAE v5.0., and summarized by type and severity in tabular format to examine their frequency, organ systems affected, severity, and relationship to study treatment.
Local control (LC) | Up to 2 years
  Defined as stable disease, partial response, or complete response based on serial imaging with CT scan. Recurrence will be defined as a suspicious mass at the site of SABR treated lesion, progressing in size on 2 consecutive computed tomography scans at a minimum interval of 1 month, combined with a positive FDG-PET defined by a SUV max ≥ 5, or a biopsy-proven confirmation.
Progression-free survival (PFS) | Up to 2 years
  Regional or distant disease progression according to RECIST v1.1 or death due to any cause
Overall survival (OS) | Up to 2 years
  A subject will be classified as either alive or dead due to any cause. The time to event will be calculated as the time from Day 1 until date of death. Day 1 is the date of 1st treatment with SABR.
Quality of life assessment | Up to 2 years
  Assessed with the Functional Assessment of Cancer Therapy: General (FACT-G)

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China